CLINICAL TRIAL: NCT00163228
Title: Functional Evaluation of Total Knee Arthroplasties,Protocol for Rising From a Chair.
Brief Title: Functional Evaluation of the Total Knee Prostheses:Rising From a Chair
Status: Withdrawn | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Johnson & Johnson (Industry)
Other Study IDs: FWB Stratec 96856; FBW Stratec 96856
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: C05.550.114.606.500; C05.550.114.606.508
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
In this study, a functional evaluation of total knee arthroplasty (TKA) patients is performed. The patients are measured prior to surgery and 6 and 12 months after surgery. The measurements consist of questionnaires and rising from a chair. Also, two types of TKA are functionally evaluated. At last, the TKA group will be compared to a THP group.

ELIGIBILITY:
Inclusion Criteria:

* unilateral TKA

Exclusion Criteria:

* TKA bilateral
* recent THP
* movement disorders like Parkinson's disease, insults, that disturb equilibrium and movements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2001-01; Study Completion 2007-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nico Verdonschot, Phd, Study Chair — ORL, Radboud University Nijmegen Medical Center; Maarten de Waal Malefijt, MD, Study Chair — ORL, Radboud University Medical Centre
Locations (1):
- ORL, Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Boonstra MC, Schreurs BW, Verdonschot N. The sit-to-stand movement: differences in performance between patients after primary total hip arthroplasty and revision total hip arthroplasty with acetabular bone impaction grafting. Phys Ther. 2011 Apr;91(4):547-54. doi: 10.2522/ptj.20090376. Epub 2011 Feb 24. PMID 21350030
- [Derived] Boonstra MC, Schwering PJ, De Waal Malefijt MC, Verdonschot N. Sit-to-stand movement as a performance-based measure for patients with total knee arthroplasty. Phys Ther. 2010 Feb;90(2):149-56. doi: 10.2522/ptj.20090119. Epub 2009 Dec 10. PMID 20007664